CLINICAL TRIAL: NCT00003639
Title: Randomised Controlled Trial of CID (Chlorambucil, Idarubicin, Dexamethasone) Versus CD (Chlorambucil, Dexamethasone) for Induction of Remission in Low Grade Non-Hodgkin's Lymphoma (Kiel Classification) Followed by Randomised Controlled Assessment of Standard Dose Interferon Versus Low Dose Interferon Versus No Further Therapy as Maintenance Treatment After Remission Induction
Brief Title: Combination Chemotherapy With or Without Interferon Alfa in Treating Patients With Low-Grade Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scotland and Newcastle Lymphoma Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066724; SNLG-NHL-VIII; EU-98034
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-05

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Interferon-alpha; Chlorambucil; Dexamethasone; Idarubicin

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: chlorambucil
Drug: dexamethasone
Drug: idarubicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells and slow the growth of non-Hodgkin's lymphoma. It is not yet known whether combining more than one chemotherapy drug with interferon alfa is more effective than chemotherapy alone in treating patients with low-grade non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without interferon alfa in treating patients with low-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the remission induction rates and toxicity of chlorambucil plus dexamethasone with or without idarubicin in patients with stage II-IV low grade non-Hodgkin's lymphoma. II. Assess the additional value of a period of consolidation/maintenance treatment utilizing low dose interferon alfa or standard dose interferon alfa versus no further treatment in relationship to the duration of event-free survival in these patients.

OUTLINE: This is a randomized, open label, controlled, multicenter study. Patients are randomized into one of two arms for induction chemotherapy. Arm I: Patients receive oral chlorambucil three times daily for 3 consecutive days, oral idarubicin daily for 3 consecutive days, and oral dexamethasone twice daily for 5 consecutive days every 21 days. Arm II: Patients receive oral chlorambucil three times daily for 3 consecutive days and oral dexamethasone twice daily for 5 consecutive days every 21 days. Treatment for both arms continues for up to 6 courses in the absence of disease progression or unacceptable toxicity. After 6 courses of chemotherapy, patients are reassessed. If they have achieved maximal complete response or good partial response, patients are randomized into one of three arms. Arm I: Patients receive no further treatment until disease progresses. Arm II: Patients receive low dose interferon alfa subcutaneously three times per week for a maximum of 3 years in the absence of disease progression. Arm III: Patients receive standard dose interferon alfa subcutaneously three times a week for a maximum of 3 years in the absence of disease progression. Patients are followed every 8-12 weeks for 3 years.

PROJECTED ACCRUAL: There will be 200 patients accrued into this study with approximately 150 patients entering the second phase of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed B cell low grade non-Hodgkin's lymphoma Stage II, III or IV Measurable disease No chronic lymphatic leukemia, prolymphocytic leukemia and hairy cell leukemia, angioimmunoblastic lymphadenopathy, mycosis fungoides, Sezary's syndrome and T-zone lymphoma, plasmacytoma, T cell lymphomas, or centroblastic lymphoma No CNS disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 15 to 70 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 2,000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.96 mg/dL AST/ALT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.65 mg/dL OR Creatinine clearance no greater than 40 mL/min Cardiovascular: No history of myocardial infarction in the past 12 months No severe or uncontrolled cardiac failure Other: No history of malignant disease except basal cell carcinoma or carcinoma in situ of the cervix No active peptic ulceration, significant dyspepsia, or history of hematemesis or melena No concurrent medical or psychological condition that may preclude study participation Not pregnant Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior extensive radiotherapy for any malignant disease Prior radiotherapy for localized disease that subsequently relapses permitted Surgery: Not specified

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1993-11

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Proctor, MD, FRCP, FRCPath, Study Chair — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Royal Victoria Infirmary, Newcastle upon Tyne, England, United Kingdom